CLINICAL TRIAL: NCT03182894
Title: A Phase IB/II Study of Epacadostat (INCB024360) in Combination With Pembrolizumab (MK-3475) and Azacitidine in Subjects With Chemo-refractory Metastatic Colorectal Cancer
Brief Title: Epacadostat in Combination With Pembrolizumab and Azacitidine in Subjects With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study will not be conducted due to changes related to the investigational agent.
Sponsor: James J Lee (Other)
Collaborators: Incyte Corporation (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, James J Lee, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 16-123
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: chemo-refractory; pembrolizumab; epacadostat; azacitidine; recommended phase 2 dose (RP2D); microsatellite-stable (MSS) Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Spinocerebellar Degenerations | interventions — epacadostat; pembrolizumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epacadostat + Pembrolizumab + Azacitidine (Experimental): Oral Epacadostat (INCB024360) (50, 100, or 300 mg twice per day,on days 1-21 of each cycle, every 21 days) in combination with Pembrolizumab (MK-3475) (200 mg IV on days 1 of each cycle, every 21 days) and Azacitidine (VIDAZA) (100 mg SQ daily on days 1-5 of each cycle, every 21 days)
  Interventions: Drug: Epacadostat (INCB024360) in Combination with Pembrolizumab (MK-3475) and Azacitidine (VIDAZA)

INTERVENTIONS:
Drug: Epacadostat (INCB024360) in Combination with Pembrolizumab (MK-3475) and Azacitidine (VIDAZA) — Oral Epacadostat (INCB024360) (50, 100, or 300 mg twice per day,on days 1-21 of each cycle, every 21 days) in combination with Pembrolizumab (MK-3475) (200 mg IV on days 1 of each cycle, every 21 days) and Azacitidine (VIDAZA) (100 mg SQ daily on days 1-5 of each cycle, every 21 days)

SUMMARY:
Trial Design This is an open label, single-arm, phase IB/II trial to evaluate the safety, tolerability and anti-tumor efficacy of epacadostat (INCB024360) in combination with pembrolizumab (MK-3475) plus azacitidine in patients with chemo-refractory MSS mCRC.

The phase 1B portion of the study will evaluate the safety, tolerability and RP2D of epacadostat (INCB024360) in combination with pembrolizumab plus azacitidine in subjects with chemo-refractory MSS mCRC without any further standard treatment options.

The phase 2 portion of the study will evaluate the efficacy and safety of epacadostat (INCB024360) in combination with pembrolizumab plus azacitidine in subjects with chemo-refractory MSS mCRC without any further standard treatment options.

In both phase IB and phase 2 portions, patients will receive the combination of azacitidine, pembrolizumab and epacadostat (INCB024360) for the first 18 cycles (Cycles 1-18). Beginning with Cycle 19 through Cycle 35, patients will receive the combination of pembrolizumab and epacadostat (INCB024360).

DETAILED DESCRIPTION:
Phase lB Portion:

* The phase 1 portion of this study will be a standard "3+3" design.
* Pembrolizumab will be administered at 200 mg intravenously (IV) on day 1 of each cycle, every 21 days.
* Azacitidine will be administered at 100 mg subcutaneous injection (SQ) daily on days 1-5 of each cycle, every 21 days
* Three dose levels of epacadostat (INCB024360) will be explored: dose levels -1, 1 and 2.
* The dose level 1 will be the starting dose level.
* If the dose level 2 is tolerable without dose limiting toxicities (DLTs), the dose level 2 will be considered the RP2D, and the phase II part will be initiated.
* DLT will be monitored during the first 21 days (cycles 1) and will be used for purposes of dose escalation and determination of RP2D.
* Definition of DLT:

Hematologic Toxicities:

* Any Grade 4 thrombocytopenia or neutropenia lasting > 7 days
* Any Grade 3 thrombocytopenia with severe bleeding

Nonhematologic Toxicities:

o Any Grade 4 toxicity EXCLUDING: Grade 4 abnormal laboratory values with a clear alternative explanation or transient (≤ 72 hours), or without associated clinically significant signs or symptoms based on investigator determination.

* Any Grade 3 or 4 AST, ALT, or total bilirubin elevation
* Any other Grade 3 toxicity EXCLUDING:

  * Nausea/vomiting controlled by medical intervention within 72 hours
  * Grade 3 rash in the absence of desquamation, no mucosal involvement, does not require systemic steroids, and resolves to Grade 1 within 14 days.
  * Grade 3 abnormal laboratory values with a clear alternative explanation or transient (≤ 72 hours), or without associated clinically significant signs or symptoms based on investigator determination.

Phase ll portion:

The phase 2 portion of this study is a non-randomized, open-label, single-arm phase II study. The primary objective of this study is to evaluate objective response rate (ORR) using RECIST1.1.

Study Procedure

* One cycle of therapy is defined as 21 days.
* Subjects may continue treatment up to 35 cycles of the study therapy (the combination of azacitidine, pembrolizumab and epacadostat [INCB024360] for the first 18 cycles [Cycle 1 to Cycle 18], and the combination of pembrolizumab and epacadostat (INCB024360) for the remaining 17 cycles [Cycle 19 to Cycle 35]) until evidence of progression of disease (PD) or unacceptable toxicity.
* Dose-limiting toxicity (DLT) will be assessed during the first 21 days (cycle 1).
* Tumor response will be determined by radiologic measurements by CT and by using RECIST. Assessment of tumor response will be performed every 3 cycles (approximately 9 weeks).
* All patients will be evaluated and graded for adverse events according to the NCI Common Terminology for Adverse Events, version 4.0 (NCI-CTCAE).

Study Treatment

* Pembrolizumab 200 mg will be administered intravenously over 30 minutes on days 1 of each cycle every 21 days.
* Azacitidine 100 mg will be administered as subcutaneous injection on days 1-5 of each cycle every 21 days.
* Epacadostat (INCB024360) will be administered orally twice a day continuously on days 1-21 of each cycle every 21 days. Two dose levels of epacadostat (INCB024360) will be explored: 100 mg BID and 300 mg BID.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be at least 18 years of age on day of signing informed consent.
3. The diagnosis of microsatellite-stable (MSS) mCRC will be based on histologic or cytologic confirmation. The histologic or cytologic confirmation of MSS status will be based on CLIA-certified immunohistochemistry (IHC) or PCR assay.
4. Have mCRC that has been previously treated with currently approved standard therapies, including fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF therapy, and, if KRAS wild type, an anti-EGFR therapy.
5. Have measurable disease based on RECIST1.1.
6. At least 1 of the tumor sites must be amenable to core needle biopsy and this may not be the site of disease used to measure antitumor response.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Life expectancy of at least 12 weeks.
9. Demonstrate adequate organ function as defined in Table 1 (Section 3.1.9), all screening labs should be performed within 14 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. Male subjects of childbearing potential (Section 5.7.2) must agree to use an adequate method of contraception as outlined in Section 5.7.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has extensive metastatic tumor burden in the liver (> 30% of liver volume) with serum albumin <3.0 g/dL.
7. Has known renal tubular acidosis with serum bicarbonate <20 mEq/L.
8. Has a known hypersensitivity to azacitidine or mannitol.
9. Has a known history of active TB (Bacillus Tuberculosis)
10. Hypersensitivity to pembrolizumab or epacadostat (INCB024360) or any of their excipients.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
14. Has an active infection requiring systemic therapy.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
18. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways), or indoleamine 2,3-dioxygenase (IDO) inhibitor.
19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
21. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

    Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
22. Any history of serotonin syndrome after receiving 1 or more serotonergic drugs.
23. Use of any monoamine oxidase inhibitor (MAOI) or drug associated with significant monoamine oxidase (MAO) inhibitory activity (listed in Tabel 4; Section 5.5) within 21 days of cycle 1 day 1.
24. Use of any melatonin supplements within 21 days of cycle 1 day 1.
25. Use of any UGT1A9 inhibitor, including (Section 5.5): acitretin, amitriptyline, androsterone, cyclosporine, dasatinib, diclofenac, diflunisal, efavirenz, erlotinib, estradiol (17-beta), flutamide, geftinib, gemfibrozil, glycyrrhetinic acid glycyrrhizin, imatinib, imipramine, ketoconazole, linoleic acid, mefenamic acid, mycophenolic acid, niflumic acid, nilotinib, phenobarbital, phenylbutazone, phenytoin, probenecid, propofol, quinidine, ritonavir, Sorafenib, sulfinpyrazone, valproic acid, and verapamil within 21 days of cycle 1 day 1.

    Note: Propofol, when used for short-term sedation during surgical/biopsy procedures, is allowed after consultation with the protocol chair or sponsor. Please check the detailed instruction for the use of propofol in Section 5.5)
26. Presence of a gastrointestinal condition that may affect drug absorption.
27. History or presence of an abnormal electrocardiogram (ECG) which, in the investigator's opinion, is clinically meaningful. Subjects with screening QTc interval > 480 ms are excluded. For subjects with an intraventricular conduction delay (QRS interval 120 ms), the JTc interval may be used in place of the QTc with sponsor approval. Subjects with left bundle branch block are excluded. Subjects with QTc prolongation due to a pacemaker may enroll if the JT is normal or with medical monitor approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase lB: Recommended phase 2 dose (RP2D) of epacadostat (INCB024360) plus pembrolizumab plus azacitidine | Up to 12 months
  Recommended phase 2 dose (RP2D) of epacadostat (INCB024360) in combination with pembrolizumab plus azacitidine in subjects with chemo-refractory microsatellite-stable (MSS) mCRC without any further standard treatment options.
Phase ll: Objective Response Rate (ORR) | Up to 18 months
  The proportion of patients with the best response of complete response (CR), or partial response (PR) by RECIST1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 18 months
  The number of months from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression).
Duration of response (DoR) | Up to 18 months
  The number of months from the date of first response (complete response (CR) or partial response (PR)) until the date of first documented disease progression or death.
Overall survival (OS) | Up to 18 months
  The number of months from the initial date of treatment to the recorded date of death.

CONTACTS AND LOCATIONS:
Overall Officials: James J Lee, MD, PhD, Study Chair — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No